CLINICAL TRIAL: NCT06560918
Title: Self-efficacy-based Auditory Rehabilitation to Optimize Real-world Outcomes With Over-the-Counter Hearing Aids: A Pilot Study
Brief Title: Self-efficacy-based Auditory Rehabilitation With Over-the-Counter Hearing Aids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 297731
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-post single arm design (Experimental): Participants will wear the hearing aids for a week while receiving the SEBAR. Outcomes will be assessed with and without hearing aids.
  Interventions: Device: hearing aids

INTERVENTIONS:
Device: hearing aids — OTC devices for a week

SUMMARY:
This goal of this study is to learn if a new audiology treatment process called the self-efficacy-based auditory rehabilitation (SEBAR) can improve confidence and success with over-the-counter (OTC) hearing aids.

The main questions it aims to answer are:

* Can the SEBAR improve participants' confidence related to managing their over-the-counter hearing aids?
* Can the SEBAR improve participants' willingness to adopt over-the-counter hearing aids, their satisfaction, quality of life, and their emotional state? Researchers will compare these outcomes of the SEBAR with and without wearing OTC hearing aids.

Participants will:

* Visit for one appointment to complete a few questionnaires without OTC hearing aids
* Wear a pair of ITC hearing aids for a week and use an app to answer questions about their experiences
* Visit for a second appointment to complete the same questionnaires with OTC hearing aids.

DETAILED DESCRIPTION:
The proposed study will use a single-arm pre-post intervention research design to achieve both the aims. Participants will complete two appointments. Assessments in the first appointment will serve as the baseline (unaided). This will be followed by a week of OTC HA use and SEBAR implementation in their natural listening situations and the outcome measures will be completed again in appointment 2 (aided) to reflect the impact of wearing OTC HAs. Scores on the outcome measures will be compared between the unaided and the aided conditions to answer both the aims. Both the appointments in the proposed study will be completed in the shared and dedicated research spaces in the Department of Audiology and Speech Pathology, College of Health Professions at the University of Arkansas for Medical Sciences. The research proposal will be submitted for the university's Institutional Review Board's approval Upon arrival participants will complete the consent process in which the PI will describe in detail all study procedures, risks and benefits of the study, and the lack of negative consequences should the participant choose to withdraw from the study or cease participation during data collection. Once the consent form has been signed, the participant will complete two appointments.

Appointment 1: For each interested participant, a standard audiometric procedure will be completed to confirm their eligibility. Once the eligible participants consent, preliminary measures will be completed. Participants will then complete the unaided baseline outcome measures of hearing aid self-efficacy, willingness to adopt HAs, expected HA satisfaction, current emotional state, and quality of life. At this time, OTC HAs will be fitted to the participants and they will receive the SEBAR. Participants will be instructed to use the HAs for at least 4 hours every day for the next week. Finally, the EMA app will be installed on their phone and its use at home will be demonstrated by the researcher.

Appointment 2: At this appointment, data from the EMA app during the one-week field trial will be stored. HAs will be tested using the Verifit 2 to verify if they are providing the required amount of amplification at the participants' preferred settings. All the outcome measures conducted will be repeated to reflect the outcomes after using the OTC HAs for a week.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 - 85 years old

  * Non-fluctuating, adult-onset, bilateral mild-to-moderate sensorineural hearing loss (average hearing thresholds for 500-3000Hz between 25- and 60-dB HL and no more than 10 dB difference between ears).
  * No previous experience with hearing aids
  * English as their first language with good self-reported health

Exclusion Criteria:

* Any reported history of outer or middle ear pathologies • No participants will be excluded based on their gender, race/ethnicity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Hearing Aid Self-Efficacy | 1 week
  Measured in unaided and aided condition

SECONDARY OUTCOMES:
Willingness to adopt hearing aids | 1 week
  Their readiness for adoption using the modified URICA
hearing aid satisfaction | 1 week
  using the SADL
emotional state | 1 week
  in the unaided and aided condition using the PANAS-SF
Hearing-related Quality of Life | 1 week
  Using one-question reflecting degree of change in quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Audiology, University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No